CLINICAL TRIAL: NCT02908243
Title: Outcomes of Prophylaxis and On-demand Treatment for Severe Hemophiliacs and Collection of Baseline Data in Hemophiliacs in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taiwan Society of Thrombosis and Hemostasis (Other)
Collaborators: Changhua Christian Hospital (Other); Taipei Medical University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taipei Medical University Shuang Ho Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 141115
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Hemophilia
Keywords: Hemophilia; Primary prophylaxis; Pettersson Score; Joint function study; Comorbidity
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Prophylaxis: Severe hemophilia A patients who receive factor VIII with dose of 15-25 IU/Kg, 2-3 times/week Severe hemophilia B patients who receive factor IX with dose of 30-50 IU/Kg, 1-2 times/week
- On-demand: Severe hemophilia A patients who receive factor VIII injection when bleeding occurs with the dose according to the criteria of World Federation of Hemophilia (WFH); Severe hemophilia B patients who receive factor IX injection when bleeding occurs with the dose according to the criteria of World Federation of Hemophilia (WFH)
- Collection of baseline data in all hemophilia A and B patients: All severe, moderate and mild types of hemophilia A and B patients
  Interventions: Other: collection of baseline data

INTERVENTIONS:
Other: collection of baseline data — collection of baseline data including ages, types, severity, inhibitors and comorbidities
  Groups: Collection of baseline data in all hemophilia A and B patients

SUMMARY:
Primary prophylaxis in severe hemophiliacs is defined that prophylaxis therapy starts before 2 years of age and prior to any clinically evident joint bleeding or after first joint bleeding and prior to the onset of joint damage irrespective of age, joints can be kept normal or very mildly damaged till teenage or adulthood. Primary prophylaxis has been proved to be more beneficial and cause less damage to joint than "on-demand" therapy. Primary prophylaxis is also known to be able to decrease the occurrence of factor VIII inhibitor and is the most advanced and useful, cost-effective therapy for hemophilia care. However, it requires 2 to 3 injections of factor VIII or IX of 20-50 IU/Kg doses every week, it costs a lot of expenses. In the year 2013, we tried hard to discuss with Bureau of National Health Insurance (BNHI) and have meeting a couple of time, eventually a guideline of an intermediate-dose prophylaxis for severe hemophilia was established and a consensus was reached that this prophylactic treatment will be cost effective without increased burden of total budget. This guideline was finally approved by BNHI and will be implemented from July 1st, 2014. In oder to evaluate the efficacy of prophylaxis treatment, patients will be arranged to come back to each hemophilia center at least once a year to have investigation of doses and annual consumption of clotting factors, frequencies and causes of bleedings, especially joint bleedings, joint outcome by studies of hemophilia joint health score (HJHS), hemophilia actives list and health-related quality of life. These results will be collected and compared between intermediate-dose prophylaxis group of patients and on demand treatment group of patients.

The life span of hemophiliacs has been improved remarkably in recent years due to sufficient and adequate treatments, especially prophylaxis treatment, therefore comorbidities in the hemophilic population, e.g. hypertension, diabetes, hyperlipidemia and cancer, etc, have been found with prevalences close to those in non-hemophilic population. It is worth that the prevalence of these comorbidity will also be investigated. In addition, basic data of the patients including age, sex, severity, the development of inhibitor and viral infection etc will also be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* all severe hemophilia A and B patients more than 2 years of age and without inhibitor

Exclusion Criteria:

* female hemophilia
* hemophiliac patients with inhibitor > = 0.6 Bethesda unit (BU)

Ages: 2 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 Severe hemophilia A patients
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
annual bleeding rate | through study completion, an average of 1 year
  spontaneous and traumatic joint and other site bleedings

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ching Shen, BS, Study Chair — Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Plan to share whole data